CLINICAL TRIAL: NCT02718248
Title: Pilot Study of a Smart Phone Assisted Problem Solving Therapy for Men Who Have Presented With Intentional Self-harm to Emergency Departments
Brief Title: Ottawa Suicide Prevention in Men Pilot Study
Acronym: OSSUPilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ottawa (Other)
Responsible Party: Principal Investigator, Dr. Simon Hatcher, Vice Chair of Research, Department of Psychiatry, University of Ottawa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20150765-01H
Record Dates: First submitted 2015-12-10; First posted 2016-03-24 (Estimated); Results first posted 2018-08-20 (Actual); Last update posted 2018-08-20 (Actual); Status verified 2017-11

CONDITIONS: Suicide
Keywords: self-harm; problem-solving therapy; emergency department; e-therapy; suicide prevention
MeSH Terms: conditions — Suicide; Self-Injurious Behavior; Emergencies; Suicide Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CHESS Mobile Health Group (Experimental): The intervention will be six weekly one hour sessions of face-to-face problem solving therapy combined with the CHESS Mobile Health smart phone application (Comprehensive Health Enhancement Support System - CHESS). The CHESS Mobile Health smart phone application enables users to access relevant resources, create a support network and check in regularly with carers. The intervention will be delivered by Dr. Hatcher, a staff psychiatrist in Liaison Psychiatry at The Ottawa Hospital General Campus.
  Interventions: Device: CHESS Mobile Health smart phone application; Behavioral: Problem solving therapy

INTERVENTIONS:
Device: CHESS Mobile Health smart phone application — A smart phone application designed to reduce intentional self-harm through problem solving e-therapy.
  Other Names: Addictions Comprehensive Health Enhancement Support System; Comprehensive Health Enhancement Support System
Behavioral: Problem solving therapy — Face to face problem solving therapy every week for six weeks.

SUMMARY:
To refine a novel intervention using a combination of a smart phone application with best practice psychotherapy for men who have presented to hospital with intentional self-harm. The outcome will be change in baseline of scores on a depression rating scale the PHQ-9 at six weeks. Moreover, the investigators will ask participants about the acceptability of the intervention and the acceptability of using routine data sources as outcome measures. This will inform methods of recruitment for the larger cluster randomized controlled trial and the creation of a treatment manual.

DETAILED DESCRIPTION:
Self-harm is defined as intentional self-poisoning or self-injury, whether or not there is evidence that the act was intended to result in death. In the past, the term used was 'attempted suicide.' However, peoples' motives for harming themselves are highly variable, a person may have more than one motive and motivation is hard to assess. In line with usual public policy in health and social care, the investigators use the term 'self-harm' describing a behaviour - avoiding the word 'deliberate' because many service users or consumers dislike its connotations.

In Ontario, the number of people who present to hospital emergency departments with self-harm is difficult to accurately assess, but the best estimate is about 30,000 each year. The most common form of self-harm seen in emergency departments (around 80% of episodes) is the intentional consumption of an excess of a medicinal or toxic product, whether or not there is evidence that the act was intended to result in death. Injuries, most commonly self-cutting, form 15-20% of episodes.

Two-thirds of people attending emergency departments because of self-harm are under 35 years of age. They are high users of health and social care services. Self-harm has a strong association with suicide: 7 patients per 1000 (about 1%) die by suicide in the year after attending emergency departments with a non-fatal episode (60 times the general population risk), rising to as many as 30 patients per 1000 over the next 15 years. In a recent longitudinal study conducted at the University of Toronto, "all-cause mortality following a first episode of self-poisoning was 1107 per 100,000 person-years… [with] nearly half of all deaths being suicides, accidents or undetermined intent." About a quarter of suicides are preceded by a hospital visit due to non-fatal self-harm in the previous year. It is the major identifiable risk factor for suicide. Mortality from non-suicidal causes is also high, with significantly more than the expected numbers of deaths from natural causes and from accidents. Whilst four of ten people who present with self-harm are men, they form nearly two thirds of suicides after an episode and are far more likely than women to die of premature death from other causes. The premature deaths are greatly over-represented among young people and the life years lost to the community are many.

Repetition of non-fatal self-harm stands at around 20% annually and is associated with much distress and many unresolved interpersonal problems. It is likely that any reduction in repetition of self-harm will be mirrored by a fall in subsequent suicides. The Canadian Association for Suicide Prevention blueprint for a National Suicide Prevention Strategy (CASP) has identified those who have presented to hospital with non-fatal self-harm as a high risk target group to reduce suicide.

People attending emergency departments after self-harm receive a variable standard of care in Ontario. Many are not assessed for psychological needs, and the little psychological therapy available is not usually covered by Ontario Health Insurance (OHIP). Local data from hospitals in Ottawa show that only 4 out of 10 men who present with intentional self-harm are seen by a mental health professional. Few are offered an evidence-based treatment aimed at reducing their risk of suicide or repeated self-harm. At present, assessment for self-harm in adults in Ontario is highly variable and there is no standard protocol for therapy. Assessment of suicide risk is currently a Required Operating Practice for Canadian Hospital accreditation; however, individuals identified as at-risk for suicide rarely receive recommended care.

Specialist services offer intensive and lengthy treatment for the minority of people who self-harm diagnosed with personality disorders, such as dialectical behavior therapy or mindfulness based therapy. The evidence for the effectiveness of these specialist therapies comes almost entirely from studies in women.

The investigators have received funding for a multicentre cluster randomized trial from the Ontario Strategy for Patient Oriented Research (SPOR) Support for People and Patient Oriented Research and Trials (SUPPORT) Unit funded by Canadian Institutes for Health Research (CIHR) and the Ontario Ministries of Health and Research and Innovation (MRI) comparing the delivery of smart phone assisted problem solving therapy with treatment as usual in men who present with self-harm. The rationale for focusing on men is that most suicides are in men and previous trials have found that providing generic treatments to everyone does not work. The intervention will build on previous work by trying to extend the range and intensity of therapy. The investigators will do this by supplementing it with a sophisticated smart phone application that has already demonstrated its effectiveness in men with substance abuse disorders. The investigators will be offering an intervention specifically designed for men who self-harm, as they are hard to engage and are more likely than women to have substance abuse problems. However, before proceeding with the full trial, a pilot study will be implemented to refine the intervention and treatment manual, as well as to test the acceptability and feasibility of the intervention to patients.

The pilot study has two aims. The first is to refine a novel intervention using a combination of a smart phone application with best practice psychotherapy for men who have presented to hospital with intentional self-harm. The primary outcome will be the change from baseline in scores on a depression rating scale the PHQ-9 at six weeks. The second aim is to test acceptability. The investigators will ask patients about the acceptability of the intervention and the acceptability of using routine data sources as outcome measures. This will inform methods of recruitment for the larger cluster randomized controlled trial. We will also create a treatment manual for problem solving therapy that incorporates the use of a smart phone application.

ELIGIBILITY:
Inclusion Criteria:

* Participant is male;
* Participant is 18 years of age or older;
* Participant has presented via Emergency Department to The Ottawa Hospital General and Civic Campuses with intentional self-harm;
* Participant is willing to return to the The Ottawa Hospital General Campus for follow-up appointments;
* Participant is willing to consent to participate in the study.

Exclusion Criteria:

* Participant is unable to read or understand English;
* Participant has cognitive impairments that render them incapable of using a smart phone;
* Participant does not have a smart phone and/or a smart phone with a data plan;
* Participants who in the opinion of the investigator will be unlikely to commit to a three month long study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Simon Hatcher, MD, PhD, Principal Investigator — University of Ottawa
Locations (2):
- Canada (2):
  - The Ottawa Hospital - General Campus, Ottawa, Ontario
  - The Ottawa Hospital - Civic Campus, Ottawa, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Canadian Institute for Health Information (2011) Health Indicators 2011. Canadian Institute for Health Information,, Ottawa, Ontario
- [Background] Hawton K, Bergen H, Casey D, Simkin S, Palmer B, Cooper J, Kapur N, Horrocks J, House A, Lilley R, Noble R, Owens D. Self-harm in England: a tale of three cities. Multicentre study of self-harm. Soc Psychiatry Psychiatr Epidemiol. 2007 Jul;42(7):513-21. doi: 10.1007/s00127-007-0199-7. Epub 2007 May 21. PMID 17516016
- [Background] Owens D, Horrocks J, House A. Fatal and non-fatal repetition of self-harm. Systematic review. Br J Psychiatry. 2002 Sep;181:193-9. doi: 10.1192/bjp.181.3.193. PMID 12204922
- [Background] Finkelstein Y, Macdonald EM, Hollands S, Sivilotti ML, Hutson JR, Mamdani MM, Koren G, Juurlink DN; Canadian Drug Safety and Effectiveness Research Network (CDSERN). Risk of Suicide Following Deliberate Self-poisoning. JAMA Psychiatry. 2015 Jun;72(6):570-5. doi: 10.1001/jamapsychiatry.2014.3188. PMID 25830811
- [Background] Da Cruz D, Pearson A, Saini P, Miles C, While D, Swinson N, Williams A, Shaw J, Appleby L, Kapur N. Emergency department contact prior to suicide in mental health patients. Emerg Med J. 2011 Jun;28(6):467-71. doi: 10.1136/emj.2009.081869. Epub 2010 Jul 26. PMID 20660941
- [Background] Hawton K, Harriss L, Zahl D. Deaths from all causes in a long-term follow-up study of 11,583 deliberate self-harm patients. Psychol Med. 2006 Mar;36(3):397-405. doi: 10.1017/S0033291705006914. Epub 2006 Jan 10. PMID 16403244
- [Background] Caterino JM, Sullivan AF, Betz ME, Espinola JA, Miller I, Camargo CA Jr, Boudreaux ED; Emergency Department Safety Assessment and Follow-up Evaluation (ED-SAFE) Investigators. Evaluating current patterns of assessment for self-harm in emergency departments: a multicenter study. Acad Emerg Med. 2013 Aug;20(8):807-15. doi: 10.1111/acem.12188. PMID 24033624
- [Background] Hawton K, Arensman E, Townsend E, Bremner S, Feldman E, Goldney R, Gunnell D, Hazell P, van Heeringen K, House A, Owens D, Sakinofsky I, Traskman-Bendz L. Deliberate self harm: systematic review of efficacy of psychosocial and pharmacological treatments in preventing repetition. BMJ. 1998 Aug 15;317(7156):441-7. doi: 10.1136/bmj.317.7156.441. PMID 9703526
- [Background] Hawton K, McKeown S, Day A, Martin P, O'Connor M, Yule J. Evaluation of out-patient counselling compared with general practitioner care following overdoses. Psychol Med. 1987 Aug;17(3):751-61. doi: 10.1017/s0033291700025988. PMID 2819914
- [Background] National Institute for Health and Clinical Excellence (2011) Longer-term care and treatment of self-harm. vol CG133.
- [Background] Carroll R, Metcalfe C, Gunnell D. Hospital management of self-harm patients and risk of repetition: systematic review and meta-analysis. J Affect Disord. 2014 Oct;168:476-83. doi: 10.1016/j.jad.2014.06.027. Epub 2014 Jun 21. PMID 25128754
- [Background] Hatcher S, Sharon C, Parag V, Collins N. Problem-solving therapy for people who present to hospital with self-harm: Zelen randomised controlled trial. Br J Psychiatry. 2011 Oct;199(4):310-6. doi: 10.1192/bjp.bp.110.090126. Epub 2011 Aug 4. PMID 21816868
- [Background] Hatcher S, Sharon C, House A, Collins N, Collings S, Pillai A. The ACCESS study: Zelen randomised controlled trial of a package of care for people presenting to hospital after self-harm. Br J Psychiatry. 2015 Mar;206(3):229-36. doi: 10.1192/bjp.bp.113.135780. Epub 2015 Jan 22. PMID 25614531
- [Background] Hatcher S, Coupe N, Durie M, Elder H, Tapsell R, Wikiriwhi K, Parag V. Te Ira Tangata: a Zelen randomised controlled trial of a treatment package including problem solving therapy compared to treatment as usual in Maori who present to hospital after self harm. Trials. 2011 May 11;12:117. doi: 10.1186/1745-6215-12-117. PMID 21569300
- [Background] Gustafson DH, McTavish FM, Chih MY, Atwood AK, Johnson RA, Boyle MG, Levy MS, Driscoll H, Chisholm SM, Dillenburg L, Isham A, Shah D. A smartphone application to support recovery from alcoholism: a randomized clinical trial. JAMA Psychiatry. 2014 May;71(5):566-72. doi: 10.1001/jamapsychiatry.2013.4642. PMID 24671165
- [Background] Hsieh HF, Shannon SE. Three approaches to qualitative content analysis. Qual Health Res. 2005 Nov;15(9):1277-88. doi: 10.1177/1049732305276687. PMID 16204405
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Psychosocial interventions for self-harm in adults. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013668. doi: 10.1002/14651858.CD013668.pub2. PMID 33884617
- [Derived] Mackie C, Dunn N, MacLean S, Testa V, Heisel M, Hatcher S. A qualitative study of a blended therapy using problem solving therapy with a customised smartphone app in men who present to hospital with intentional self-harm. Evid Based Ment Health. 2017 Nov;20(4):118-122. doi: 10.1136/eb-2017-102764. Epub 2017 Oct 13. PMID 29030503

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participant recruitment took place over a 6 month period from Sept. 2016 to Feb. 2017. TOH ED staff were asked to approach participants with information about the study and refer any eligible men to the Research Coordinator. Once participants were referred to the Research Coordinator, she contacted them by telephone and scheduled a Baseline Visit.
Pre-assignment Details: No participants were excluded from this study post-enrollment.
Period: Overall Study
Arm/Group | CHESS Mobile Health Group
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | CHESS Mobile Health Group
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.43 (8.142)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 7
Severity of Depression Symptoms [Mean (Standard Deviation); unit: units on a scale] — Severity of depression symptoms was measured using the Patient Health Questionnaire (PHQ-9). This is a 9-item self-report scale which assessed the severity of depressive symptoms over the preceding 2 weeks. Total scores on this scale range from 0 to 27, with higher scores indicating more severe depression symptoms. The scores on the Patient Health Questionnaire (PHQ-9) scale should be interpreted as follows:
  0-4: Minimal Depression; 5-9: Mild Depression 10-14: Moderate Depression; 15-19: Moderately Severe Depression; 20 and Above: Severe Depression.
  units on a scale | 18.29 (5.529)
Physical Functioning [Mean (Standard Deviation); unit: units on a scale] — Physical Functioning was measured using the Physical Functioning subscale of the Medical Outcomes Survey Short Form 12 (SF-12). The SF-12 is a 12-item self-report survey that assesses general health and well-being using a total of 8 subscales. The Physical Functioning Subscale is scored using a range of 0-100, with a higher score indicating better physical functioning.
  units on a scale | 82.14 (18.898)
Physical Role Limitations [Mean (Standard Deviation); unit: units on a scale] — Physical Role Limitations was measured using the Physical Role Limitations subscale of the Medical Outcomes Survey Short Form 12 (SF-12). The SF-12 is a 12-item self-report survey that assesses general health and well-being using a total of 8 subscales. The Physical Role Limitations Subscale is scored using a range of 0-100, with a higher score indicating fewer role limitations due to physical health difficulties.
  units on a scale | 75 (23.936)
Emotional Role Limitations [Mean (Standard Deviation); unit: units on a scale] — Emotional Role Limitations was measured using the Emotional Role Limitations subscale of the Medical Outcomes Survey Short Form 12 (SF-12). The SF-12 is a 12-item self-report survey that assesses general health and well-being using a total of 8 subscales. The Emotional Role Limitations Subscale is scored using a range of 0-100, with a higher score indicating fewer role limitations due to emotional health difficulties.
  units on a scale | 26.79 (26.446)
Vitality [Mean (Standard Deviation); unit: units on a scale] — Vitality was measured using the Vitality subscale of the Medical Outcomes Survey Short Form 12 (SF-12). The SF-12 is a 12-item self-report survey that assesses general health and well-being using a total of 8 subscales. The Vitality subscale is scored using a range of 0-100, with a higher score indicating a higher degree of vitality.
  units on a scale | 25.0 (20.412)
General Health [Mean (Standard Deviation); unit: units on a scale] — General Health was measured using the General Health subscale of the Medical Outcomes Survey Short Form 12 (SF-12). The SF-12 is a 12-item self-report survey that assesses general health and well-being using a total of 8 subscales. The General Health Subscale is scored using a range of 0-100, with a higher score indicating higher levels of general health.
  units on a scale | 42.14 (29.277)
Mental Health Functioning [Mean (Standard Deviation); unit: units on a scale] — Mental Health Functioning was measured using the Mental Health subscale of the Medical Outcomes Survey Short Form 12 (SF-12). The SF-12 is a 12-item self-report survey that assesses general health and well-being using a total of 8 subscales. The Mental Health Functioning Subscale is scored using a range of 0-100, with a higher score indicating better mental health functioning.
  units on a scale | 17.86 (17.466)
Bodily Pain [Mean (Standard Deviation); unit: units on a scale] — Bodily Pain was measured using the Bodily Pain subscale of the Medical Outcomes Survey Short Form 12 (SF-12). The SF-12 is a 12-item self-report survey that assesses general health and well-being using a total of 8 subscales. The Bodily Pain Subscale is scored using a range of 0-100, with a higher score indicating lower levels of bodily pain.
  units on a scale | 71.43 (30.375)
Social Functioning [Mean (Standard Deviation); unit: units on a scale] — Social Functioning was measured using the Social Functioning subscale of the Medical Outcomes Survey Short Form 12 (SF-12). The SF-12 is a 12-item self-report survey that assesses general health and well-being using a total of 8 subscales. The Social Functioning Subscale is scored using a range of 0-100, with a higher score indicating higher social functioning.
  units on a scale | 28.57 (22.493)
General Health Related Quality of Life [Median (Full Range); unit: units on a scale] — Generic health-related quality of life index. The total scores on this measure range from 11111 to 33333, with lower values indicating higher levels of health-related quality of life.
  units on a scale | 11223 [11113 to 21223]
EuroQol 5 Dimensions Visual Analytic Scale [Mean (Standard Deviation); unit: units on a scale] — Participants were asked to use the EuroQol 5 Dimensions Visual Analytic Scale to assess their overall health on a scale from 0 to 100, with 100 being the best possible health state.
  units on a scale | 47.57 (11.530)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Scores on the Patient Health Questionnaire (PHQ-9) Scale at Week 6
Description: Measures change in the severity of depressive symptoms. Total scores on this scale range from 0 to 27, with higher scores indicating more severe depression symptoms. The scores on the Patient Health Questionnaire (PHQ-9) scale should be interpreted as follows:
  0-4: Minimal Depression; 5-9: Mild Depression 10-14: Moderate Depression; 15-19: Moderately Severe Depression; 20 and Above: Severe Depression.
Time Frame: Baseline, Week 1, Week 2, Week 3, Week 4, Week 5
Population: Throughout the course of the study, the following study time points were missed: Week 1 (2 participants), Week 3 (1 participant) and Week 4 (1 participant).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CHESS Mobile Health Group
Number analyzed (Participants) | 7
units on a scale
  Week 1: number analyzed (Participants) | 5
  Week 1 | 19.8 (5.07)
  Week 2: number analyzed (Participants) | 6
  Week 2 | 15.17 (5.565)
  Week 3 | 16.86 (6.619)
  Week 4: number analyzed (Participants) | 6
  Week 4 | 16.83 (6.853)
  Week 5 | 13.71 (9.995)

2. Secondary Outcome: Physical Functioning
Description: Physical Functioning was measured using the Physical Functioning subscale of the Medical Outcomes Survey Short Form 12 (SF-12). The SF-12 is a 12-item self-report survey that assesses general health and well-being using a total of 8 subscales. The Physical Functioning Subscale is scored using a range of 0-100, with a higher score indicating better physical functioning.
Time Frame: Baseline and Week 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CHESS Mobile Health Group
Number analyzed (Participants) | 7
units on a scale
  Baseline | 82.14 (18.898)
  Week 5 | 92.86 (18.898)

3. Secondary Outcome: Physical Role Limitations
Description: Physical Role Limitations was measured using the Physical Role Limitations subscale of the Medical Outcomes Survey Short Form 12 (SF-12). The SF-12 is a 12-item self-report survey that assesses general health and well-being using a total of 8 subscales. The Physical Role Limitations Subscale is scored using a range of 0-100, with a higher score indicating fewer role limitations due to physical health difficulties.
Time Frame: Baseline, Week 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CHESS Mobile Health Group
Number analyzed (Participants) | 7
units on a scale
  Baseline | 75.0 (23.936)
  Week 5 | 83.93 (18.70)

4. Secondary Outcome: Emotional Role Limitations
Description: Emotional Role Limitations was measured using the Emotional Role Limitations subscale of the Medical Outcomes Survey Short Form 12 (SF-12). The SF-12 is a 12-item self-report survey that assesses general health and well-being using a total of 8 subscales. The Emotional Role Limitations Subscale is scored using a range of 0-100, with a higher score indicating fewer role limitations due to emotional health difficulties.
Time Frame: Baseline, Week 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CHESS Mobile Health Group
Number analyzed (Participants) | 7
units on a scale
  Baseline | 26.79 (26.446)
  Week 5 | 44.64 (25.877)

5. Secondary Outcome: Vitality
Description: Vitality was measured using the Vitality subscale of the Medical Outcomes Survey Short Form 12 (SF-12). The SF-12 is a 12-item self-report survey that assesses general health and well-being using a total of 8 subscales. The Vitality subscale is scored using a range of 0-100, with a higher score indicating a higher degree of vitality.
Time Frame: Baseline, Week 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CHESS Mobile Health Group
Number analyzed (Participants) | 7
units on a scale
  Baseline | 25.00 (20.412)
  Week 5 | 46.43 (33.63)

6. Secondary Outcome: General Health
Description: General Health was measured using the General Health subscale of the Medical Outcomes Survey Short Form 12 (SF-12). The SF-12 is a 12-item self-report survey that assesses general health and well-being using a total of 8 subscales. The General Health Subscale is scored using a range of 0-100, with a higher score indicating higher levels of general health.
Time Frame: Baseline, Week 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CHESS Mobile Health Group
Number analyzed (Participants) | 7
units on a scale
  Baseline | 42.14 (29.277)
  Week 5 | 48.57 (23.755)

7. Secondary Outcome: Mental Health Functioning
Description: Mental Health Functioning was measured using the Mental Health subscale of the Medical Outcomes Survey Short Form 12 (SF-12). The SF-12 is a 12-item self-report survey that assesses general health and well-being using a total of 8 subscales. The Mental Health Functioning Subscale is scored using a range of 0-100, with a higher score indicating better mental health functioning.
Time Frame: Baseline, Week 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CHESS Mobile Health Group
Number analyzed (Participants) | 7
units on a scale
  Baseline | 17.86 (17.466)
  Week 5 | 30.36 (21.478)

8. Secondary Outcome: Bodily Pain
Description: Bodily Pain was measured using the Bodily Pain subscale of the Medical Outcomes Survey Short Form 12 (SF-12). The SF-12 is a 12-item self-report survey that assesses general health and well-being using a total of 8 subscales. The Bodily Pain Subscale is scored using a range of 0-100, with a higher score indicating lower levels of bodily pain.
Time Frame: Baseline, Week 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CHESS Mobile Health Group
Number analyzed (Participants) | 7
units on a scale
  Baseline | 71.43 (30.375)
  Week 5 | 82.14 (18.898)

9. Secondary Outcome: Social Functioning
Description: Social Functioning was measured using the Social Functioning subscale of the Medical Outcomes Survey Short Form 12 (SF-12). The SF-12 is a 12-item self-report survey that assesses general health and well-being using a total of 8 subscales. The Social Functioning Subscale is scored using a range of 0-100, with a higher score indicating higher social functioning.
Time Frame: Baseline, Week 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CHESS Mobile Health Group
Number analyzed (Participants) | 7
units on a scale
  Baseline | 28.57 (22.493)
  Week 5 | 35.71 (19.67)

10. Secondary Outcome: Health-Related Quality of Life
Description: Generic health-related quality of life index. The total scores on this measure range from 11111 to 33333, with lower values indicating higher levels of health-related quality of life.
Time Frame: Baseline and Week 5
Measure: Median (Full Range); unit: units on a scale
Arm/Group | CHESS Mobile Health Group
Number analyzed (Participants) | 7
units on a scale
  Baseline | 11223 [11113 to 21223]
  Week 5 | 11313 [11111 to 22223]

11. Secondary Outcome: Perceived Overall Health
Description: Participants were asked to use the EuroQol 5 Dimensions Visual Analytic Scale to assess their overall health on a scale from 0 to 100, with 100 being the best possible health state.
Time Frame: Baseline, Week 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CHESS Mobile Health Group
Number analyzed (Participants) | 7
units on a scale
  Baseline | 47.57 (11.53)
  Week 5 | 60.29 (14.795)

12. Secondary Outcome: Participant Exit Questionnaire
Description: The investigators will ask participants about the user comprehension, user practicality and the methods of data collection with regards to the CHESS Mobile Health smart phone application. The Participant Exit Questionnaire will also ask that users make comments or suggestions for future use and development of the application. This will test the acceptability of the intervention and the acceptability of using routine data sources as outcome measures.
Time Frame: within 4 months of study completion
Measure: Number; unit: percentage of participants who agreed
Arm/Group | CHESS Mobile Health Group
Number analyzed (Participants) | 7
percentage of participants who agreed
  Application Easy to Install | 100.0
  Application is User Friendly | 85.7
  Application was easy to use | 71.4
  PST is a good fit for me | 71.4
  In PST we worked on what I wanted | 85.7
  Application was useful | 28.6
  I would use the application again | 42.9

13. Other Pre Specified Outcome: Recruitment Rates at 6 Months
Description: Will be used to assess the feasibility of recruitment for a larger, multicentre cluster randomized controlled trial (RCT). To test feasibility in patients the investigators aim to recruit at least half of the men the study team ask to take part in the pilot study. To test feasibility in referring clinicians, the aim is that at least half of men who present with intentional self-harm to the psychiatric emergency service will be approached and complete the The Ottawa Hospital (TOH) form allowing contact details to be passed on to researchers.
Time Frame: Within 6 months of study launch
Population: This group includes all participants referred to the study (N=15).
Measure: Number; unit: percentage of participants enrolled
Arm/Group | CHESS Mobile Health Group
Number analyzed (Participants) | 15
percentage of participants enrolled | 46.6

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: Adverse events related to subsequent self-harm were collected from participants by their therapist at each study visit.
Arm/Group | CHESS Mobile Health Group
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 5/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CHESS Mobile Health Group (N=7)
Subsequent Self-Harm (Injury, poisoning and procedural complications) | 3 (4) — Intentional self-harm
Tooth Abscess (Infections and infestations) | 1 (1)
Trip (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-30): https://cdn.clinicaltrials.gov/large-docs/48/NCT02718248/Prot_SAP_000.pdf